CLINICAL TRIAL: NCT04288804
Title: A Study to Analyze Features of Dysphonia and Tremor in PD Patients to Aid in the Development of an Accurate Diagnostic Tool for Early-Detection of PD
Brief Title: A Study to Analyze Symptoms Prevalent in Early PD (Dysphonia, Tremor)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goalspal LLC (Other)
Responsible Party: Sponsor
Other Study IDs: NIA0117210
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Dysphonia; Tremor; Neurological Disorder; Web-based; Neurological Disease
MeSH Terms: conditions — Parkinson Disease; Dysphonia; Tremor; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Accelerometer data, voice recording, question responses (age-group, gender, PD/non-PD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control (healthy, non-PD participants): An audio file made up of a voice recording of the sustained short a vowel sound, along with accelerometer data while maintaining various positions, will be collected.
  Interventions: Device: Smartphone microphone sensor; Device: Smartphone accelerometer sensor
- PD: An audio file made up of a voice recording of the sustained short a vowel sound, along with accelerometer data while maintaining various positions, will be collected.
  Interventions: Device: Smartphone microphone sensor; Device: Smartphone accelerometer sensor

INTERVENTIONS:
Device: Smartphone microphone sensor — The volunteer will record themselves sustaining the short a vowel sound for 10 seconds.
Device: Smartphone accelerometer sensor — The volunteer's smartphone's accelerometer will record accelerometer data (positions on the x, y, and z axes) while the volunteer maintains 4 positions, each for 10 seconds.

SUMMARY:
This is a web-based study that involves monitoring hallmark symptoms of Parkinson's Disease (PD), specifically dysphonia and tremor, using smartphone sensor data. The entire length of the study will only take 5 minutes, so volunteers will not have to repeatedly contribute data. The study is made up of 5 short, 10-second long activities, which include sustaining the short a vowel sound to monitor changes in vocal fundamental frequency and holding a smartphone in different positions on either side of the body to measure changes in amplitude. To be a part of this study, volunteers must have an iPhone that is running on the software iOS 13 or higher, because they will be asked to download a smartphone application from an online App Store.

DETAILED DESCRIPTION:
Participants will be asked to complete a series of activities, as outlined below.

1. They will be asked to turn on "Do Not Disturb" and set their smartphone's volume to the maximum. This is to ensure that they can hear narrated instructions guiding them through the activities to come, and that data collection is uninterrupted.
2. Volunteers will sustain the short a vowel sound for 10 seconds. This is to analyze PD-related dysphonia.
3. Volunteers will place their smartphone in their left hand and rest it in their lap for 10 seconds. This is to analyze PD-related rest tremor on the left side of the body. (Duration: 10 seconds)
4. Volunteers will place their smartphone in their right hand and rest it in their lap for 10 seconds. This is to analyze PD-related rest tremor on the right side of the body. (Duration: 10 seconds)
5. Volunteers will hold their smartphone face-down at shoulder-level, in their left hand. This is to analyze PD-related postural tremor on the left side of the body. (Duration: 10 seconds)
6. Volunteers will hold their smartphone face-down at shoulder-level, in their right hand. This is to analyze PD-related postural tremor on the right side of the body. (Duration: 10 seconds)

Finally, participants will be asked to indicate their gender, age group, and status (whether or not they have PD), for data-labeling purposes. Please note that all data is collected anonymously and thus cannot be tracked down to a specific participant. Nevertheless, it will be encrypted and stored in a secure database, with each participant corresponding to a GUID (Global Unique Identifier), although participants will not be asked for their name. As this is not a medical study, there are no expected medical side effects, however, certain activities and questions may seem frustrating and boring.

Participants will mainly benefit from the study indirectly, as it will increase understanding of symptoms prevalent in early PD, and may contribute to the development of diagnostic tools.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease (PD)
* Healthy

Exclusion Criteria:

* Subject does not have clinical diagnosis of PD, however, has another neurological disorder/disease that manifests with symptoms of tremor or dysphonia
* Subject diagnosed with PD does not have dysphonia and tremor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects must be healthy controls, or clinically diagnosed with PD in order to participate. They also may not have another illness that causes tremor and/or dysphonia - subjects who have PD must also have PD-related dysphonia and PD-related tremor.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2023-12-26 (Estimated)

PRIMARY OUTCOMES:
PD-related Tremor | 40 seconds
  24 features, composed of mean absolute deviation and mean standard deviation for each axis (x, y, z), for 4 likely occurrences of tremor, will be observed by looking at the accelerometer data file of each participant.
PD-related Dysphonia | 10 seconds
  Features, composed of vocal fundamental frequency, and similar measures to jitter and shimmer, will be observed by looking at the mel spectrogram for the audio file of each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Goalspal LLC, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified participant data may be made available to other researchers in a compiled dataset. 24 accelerometer features from each participant will be included in their entry, tagged by a GUID. Along with this, an audio file of them sustaining the short a vowel sound for 10 seconds will be a part of their entry. Finally, their status (control/PD), gender, and age-group will be included, so that statistical analyses can be made.

REFERENCES:
- See also: A visual protocol of what the study entails, complete with pictures of each screen wherein a volunteer must complete a certain activity, and how to download the mobile study. — http://cepha.ai